CLINICAL TRIAL: NCT02881658
Title: The Effect of Soya Beverage Fortified With Plant Sterol on Major Serum Lipids in Normocholesterolemic, Healthy Southern Chinese Individuals
Brief Title: The Effect of 3-Week Consumption of Soya Beverage Enriched With Plant Sterols on Serum LDL-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Bernard Cheung, Professor of Department of Medicine, HKU, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CTC1521
Record Dates: First submitted 2016-08-14; First posted 2016-08-29 (Estimated); Results first posted 2017-09-21 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Dyslipidemia
Keywords: Plant sterols; Low-Density Lipoprotein Cholesterol; Phytosterols; Soya Beverage
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Plant sterols-enriched soya beverage provided by Vitasoy (Experimental): Daily consumption of 2g of plant sterols as provided by one pack of 250 ml of plant sterols-enriched soya beverage for consecutive 3 weeks, each pack consumed once with main meal (i.e breakfast, lunch or dinner).
  Interventions: Dietary Supplement: Plant sterols-enriched soya beverage provided by Vitasoy
- Soya beverage provided by Vitasoy (Placebo Comparator): Daily consumption of one pack of 250 ml of soya beverage (without plant sterols) for consecutive 3 weeks, each pack consumed once with main meal (i.e breakfast, lunch or dinner).
  Interventions: Dietary Supplement: Soya beverage provided by Vitasoy

INTERVENTIONS:
Dietary Supplement: Plant sterols-enriched soya beverage provided by Vitasoy — the study product is a 2g plant sterols-enriched in 250ml soya beverage
  Arms: Plant sterols-enriched soya beverage provided by Vitasoy
Dietary Supplement: Soya beverage provided by Vitasoy — the placebo product is a 250 ml soya beverage
  Arms: Soya beverage provided by Vitasoy

SUMMARY:
This is a local, single-center, two-arm, randomized, double-blind, placebo-controlled clinical trial that examines the LDL-C-lowering effect of the consumption of a soya beverage enriched with plant sterol for 3 weeks. This study also examines if there is other health-benefits by consuming the plant sterols fortified soya beverage in terms of serum total triglyceride, total and HDL cholesterol, other cardiometabolic risk factors and musculoskeletal-related traits including handgrip strength, gait speed, peak expiratory flow rate, bio-impedance and body balance.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the third commonest cause of deaths in Hong Kong and accounting for 14.4% of all deaths in 2012. Robust data attest the causal role of low-density lipoprotein cholesterol (LDL-C) in the development and progression of CVD. Reduction of LDL-C levels achieved by pharmacological agents in conjunction with diet change has been demonstrated to significantly reduce CVD morbidity and mortality. Moreover, it has been frequently reported that dietary incorporation of plant sterols/stanols could reduce blood LDL-C level in both healthy and dyslipidaemic individuals with great inter-individual variability of LDL-C response. Therefore, functional food enriched with plant sterols/stanols not only may provide additional LDL-C lowering benefit in dyslipidaemic patients as an adjunct to traditional pharmacologic therapy, but also play a role in primary prevention of CVD in the general population.

ELIGIBILITY:
Inclusion Criteria:

* Southern Chinese male or female ≥ 18 years;
* In good general health as evidenced by medical history;
* Have the ability to understand the requirements of the study, provide written informed consent, including consent for the use and disclose of research-related health information, and comply with the study data collection procedures. Provide signed and dated informed consent form

Exclusion Criteria:

* Subject with familial hypercholesterolemia;
* On regular medication(s) which affect gastrointestinal functions and blood lipids level for the past 3 months, such as, but not limited to:

  * Antibiotics of >1 week duration
  * GI related medications such as antacids
* Having blood lipid lowering medications such as statins, selective cholesterol absorption inhibitors (e.g. ezetimibe), fibrates, niacin, resins, omega- 3
* Heavy-smokers (more than 1 pack per day)
* Subject with heavy alcohol intake (>40 g/day for men ; >30 g/day for women) (32), or having history of alcohol abuse within 12 months prior to the study
* Subjects with taste aversion to placebo/intervention soya beverages
* Subject refusing to stop the consumption of plant sterols-enriched products if any during the study (other than the studied product) or having regular consumption of sterols/stanols cholesterol-lowering supplements/functional foods or other related products such as:

  * Sterol/ Stanol - containing margarines, milk, yoghurt drink and soya beverages
  * Sterol / Stanol supplements
  * Fish oils & omega-3 supplements
* Subject receiving systemic treatment or topical treatment likely to interfere with evaluation of the study parameters
* Subject currently involved in a clinical trial or in an exclusion period following participation in another clinical trial
* Pregnancy or lactation
* Having soy allergy
* Being a vegan
* Being an athlete
* Concurrently participating in weight management or dietary program
* On diet pills, such as, but not limited to chitosan and dulcolax
* With history of sitosterolemia
* Having history of hypercholesterolemia, diabetes, thyroid disease, severe kidney diseases, cardiovascular diseases, chronic gastrointestinal disorders, cancers and AIDs ( acquired immune deficiency syndrome)
* Having history of malabsorption syndrome arising from diseases such as, but not limited to celiac disease, short bowel syndrome, cystic fibrosis, pancreatitis, diseases of gall-bladder, liver or pancreas, intestinal infection, injury, surgery and radiotherapy
* Taking over-the-counter Chinese medications or supplements with cholesterol/lipid lowering and related claims
* High blood cholesterol at screening [Total cholesterol level ≥6.22mmol/L]
* High LDL cholesterol [LDL cholesterol level ≥4.15mmol/L]
* High blood triglyceride at screening [Triglyceride ≥3.39mmol/L]
* Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2016-05; Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Man Yung Cheung, Principal Investigator — Li Ka Shing Faculty of Medicine, The University of Hong Kong
Locations (1):
- Li Ka Shing Faculty of Medicine, The University of Hong Kong, Pokfulam, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Chau YP, Cheng YC, Sing CW, Tsoi MF, Cheng VK, Lee GK, Cheung CL, Cheung BMY. The lipid-lowering effect of once-daily soya drink fortified with phytosterols in normocholesterolaemic Chinese: a double-blind randomized controlled trial. Eur J Nutr. 2020 Sep;59(6):2739-2746. doi: 10.1007/s00394-019-02119-w. Epub 2019 Oct 23. PMID 31642984

RESULTS

PARTICIPANT FLOW:
Groups:
- Plant Sterols-enriched Soya Beverage Provided by Vitasoy: Daily consumption of 2g of plant sterols as provided by one pack of 250 ml of plant sterols-enriched soya beverage for consecutive 3 weeks, each pack consumed once with main meal (i.e breakfast, lunch or dinner).
  Plant sterols-enriched soya beverage: the study product is a 2g plant sterols-enriched in 250ml soya beverage
- Soya Beverage Provided by Vitasoy: Daily consumption of one pack of 250 ml of soya beverage (without plant sterols) for consecutive 3 weeks, each pack consumed once with main meal (i.e breakfast, lunch or dinner).
  Soya beverage: the placebo product is a 250 ml soya beverage
Period: Overall Study
Arm/Group | Plant Sterols-enriched Soya Beverage Provided by Vitasoy | Soya Beverage Provided by Vitasoy
Started | 100 | 101
Completed | 98 | 96
Not Completed | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Plant Sterols-enriched Soya Beverage Provided by Vitasoy | Soya Beverage Provided by Vitasoy | Total
Number analyzed (Participants) | 100 | 101 | 201
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (16.5) | 44 (16.7) | 45 (16.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 52 | 101
  Male | 51 | 49 | 100
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Mean of Serum Low-density Lipoprotein Cholesterol (LDL-C) Via Blood Test at Baseline and Week 3
Time Frame: From baseline to week 3
Population: All 201 subjects were included in the population, but certain blood test result on LDL-C were not available, thus difference in the overall number of participants analyzed and the actual number of participants included to present the mean value.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Plant Sterols-enriched Soya Beverage Provided by Vitasoy | Soya Beverage Provided by Vitasoy
Number analyzed (Participants) | 100 | 101
mmol/L
  Baseline: number analyzed (Participants) | 93 | 93
  Baseline | 2.91 (0.961) | 2.83 (0.814)
  Week 3: number analyzed (Participants) | 96 | 95
  Week 3 | 2.71 (0.830) | 2.75 (0.794)

2. Secondary Outcome: Change of Low Density Lipoprotein Cholesterol (LDL-C) Via Blood Test at Baseline and Week 3
Time Frame: From baseline to week 3
Measure: Median (Inter-Quartile Range); unit: percentage of change
Arm/Group | Plant Sterols-enriched Soya Beverage Provided by Vitasoy | Soya Beverage Provided by Vitasoy
Number analyzed (Participants) | 91 | 88
percentage of change | -7.69 [-15.36 to 2.19] | -1.56 [-10.22 to 7.43]

3. Secondary Outcome: Change of High-density Lipoprotein Cholesterol (HDL-C) Via Blood Test at Baseline and Week 3
Time Frame: From baseline to week 3
Measure: Median (Inter-Quartile Range); unit: percentage of change
Arm/Group | Plant Sterols-enriched Soya Beverage Provided by Vitasoy | Soya Beverage Provided by Vitasoy
Number analyzed (Participants) | 97 | 96
percentage of change | 0.0 [-5.56 to 7.69] | 0.0 [-6.67 to 11.11]

4. Secondary Outcome: Change of Total Cholesterol Via Blood Test at Baseline and Week 3
Time Frame: From baseline to week 3
Measure: Median (Inter-Quartile Range); unit: percentage of change
Arm/Group | Plant Sterols-enriched Soya Beverage Provided by Vitasoy | Soya Beverage Provided by Vitasoy
Number analyzed (Participants) | 97 | 96
percentage of change | -2.82 [-8.38 to 3.16] | -1.86 [-7.06 to 4.15]

5. Secondary Outcome: Change of Triglycerides (TAG) Via Blood Test at Baseline and Week 3
Time Frame: From baseline to week 3
Measure: Median (Inter-Quartile Range); unit: percentage of change
Arm/Group | Plant Sterols-enriched Soya Beverage Provided by Vitasoy | Soya Beverage Provided by Vitasoy
Number analyzed (Participants) | 97 | 96
percentage of change | 0.00 [-18.64 to 21.15] | -1.88 [-17.21 to 19.26]

6. Secondary Outcome: Change of Serum Creatinine Via Blood Test at Baseline and Week 3
Time Frame: From baseline to week 3
Measure: Median (Inter-Quartile Range); unit: percentage of change
Arm/Group | Plant Sterols-enriched Soya Beverage Provided by Vitasoy | Soya Beverage Provided by Vitasoy
Number analyzed (Participants) | 97 | 96
percentage of change | 0 [-4 to 6] | 0 [-4 to 4]

7. Secondary Outcome: Changes of Fasting Blood Glucose Via Blood Test at Baseline and Week 3
Time Frame: From baseline to week 3
Measure: Median (Inter-Quartile Range); unit: percentage of change
Arm/Group | Plant Sterols-enriched Soya Beverage Provided by Vitasoy | Soya Beverage Provided by Vitasoy
Number analyzed (Participants) | 97 | 96
percentage of change | 0.0 [-4.3 to 4.1] | 0.0 [-4.2 to 2.2]

8. Secondary Outcome: Changes of Cardiometabolic Risk Factors Via Measuring Anthropometry at Baseline and Week 3
Time Frame: From baseline to week 3
Measure: Median (Inter-Quartile Range); unit: percentage of change
Arm/Group | Plant Sterols-enriched Soya Beverage Provided by Vitasoy | Soya Beverage Provided by Vitasoy
Number analyzed (Participants) | 98 | 96
percentage of change
  Median percentage change of Body weight | -0.1 [-0.8 to 0.9] | 0.2 [-0.6 to 1.0]
  Median percentage change of Waist circumference | 0 [-2 to 3] | 0 [-3 to 3]
  Median percentage change of Hip circumference | 0 [-1 to 1] | 0 [-1 to 1]

9. Secondary Outcome: Changes of Cardiometabolic Risk Factors Via Measuring Blood Pressure at Baseline and Week 3
Time Frame: From baseline to week 3
Measure: Median (Inter-Quartile Range); unit: percentage of change
Arm/Group | Plant Sterols-enriched Soya Beverage Provided by Vitasoy | Soya Beverage Provided by Vitasoy
Number analyzed (Participants) | 98 | 96
percentage of change
  Median percentage change of Sys. blood pressure | -1 [-6 to 2] | -2 [-5 to 2]
  Median percentage change of Dia. blood pressure | -3 [-7 to 1] | -3 [-6 to 1]

10. Secondary Outcome: Changes of Cardiometabolic Risk Factors Via Measuring Body Temperature at Baseline and Week 3
Time Frame: From baseline to week 3
Measure: Median (Inter-Quartile Range); unit: percentage of body temperature change
Arm/Group | Plant Sterols-enriched Soya Beverage Provided by Vitasoy | Soya Beverage Provided by Vitasoy
Number analyzed (Participants) | 98 | 95
percentage of body temperature change | -0.3 [-0.5 to 0.0] | -0.3 [-0.5 to 0.0]

11. Secondary Outcome: Changes of Musculoskeletal-related Traits Via Measuring Hand Grip Strength at Baseline and Week 3
Time Frame: From baseline to week 3
Measure: Median (Inter-Quartile Range); unit: percentage of change
Arm/Group | Plant Sterols-enriched Soya Beverage Provided by Vitasoy | Soya Beverage Provided by Vitasoy
Number analyzed (Participants) | 92 | 95
percentage of change | 2 [-8 to 11] | 0 [-12 to 10]

12. Secondary Outcome: Changes of Musculoskeletal-related Traits Via Measuring Bio-Impedance at Baseline and Week 3
Time Frame: From baseline to week 3
Measure: Median (Inter-Quartile Range); unit: percentage of change
Arm/Group | Plant Sterols-enriched Soya Beverage Provided by Vitasoy | Soya Beverage Provided by Vitasoy
Number analyzed (Participants) | 97 | 93
percentage of change
  Median % change of Bioimpedance - Fat percentage | -1.0 [-4.1 to 1.8] | -0.8 [-3.6 to 2.1]
  Median % change of Bioimpedance - Fat mass | -1.1 [-4.8 to 2.1] | -0.7 [-3.3 to 2.9]

13. Secondary Outcome: Changes of Musculoskeletal-related Traits Via Measuring Peak Expiratory Flow Rate at Baseline and Week 3
Time Frame: From baseline to week 3
Measure: Median (Inter-Quartile Range); unit: percentage of change
Arm/Group | Plant Sterols-enriched Soya Beverage Provided by Vitasoy | Soya Beverage Provided by Vitasoy
Number analyzed (Participants) | 98 | 96
percentage of change | 0 [-5 to 7] | -0 [-5 to 6]

14. Secondary Outcome: Changes of Musculoskeletal-related Traits Via Measuring 6 Metres Gait Speed at Baseline and Week 3
Time Frame: From baseline to week 3
Measure: Median (Inter-Quartile Range); unit: percentage of change
Arm/Group | Plant Sterols-enriched Soya Beverage Provided by Vitasoy | Soya Beverage Provided by Vitasoy
Number analyzed (Participants) | 98 | 95
percentage of change | -1.74 [-7.80 to 6.81] | -1.46 [-8.41 to 9.44]

15. Secondary Outcome: Changes of Musculoskeletal-related Traits Via Measuring Centre of Pressure Excursion Index for Left and Right Foot at Baseline and Week 3
Description: centre of pressure excursion index = CPEI
Time Frame: From baseline to week 3
Measure: Median (Inter-Quartile Range); unit: Percentage of Change
Arm/Group | Plant Sterols-enriched Soya Beverage Provided by Vitasoy | Soya Beverage Provided by Vitasoy
Number analyzed (Participants) | 96 | 92
Percentage of Change
  Median percentage of CPEI change (left foot) | 0 [-22 to 26] | 0 [-21 to 24]
  Median percentage of CPEI change (right foot) | 4 [-17 to 22] | -5 [-20 to 23]

ADVERSE EVENTS:
Time Frame: Participants were asked to complete a questionnaire related to adverse event that happened during the 3 weeks period of consuming soya beverage.
Groups:
- Plant Sterols-enriched Soya Beverage: Daily consumption of 2g of plant sterols as provided by one pack of 250 ml of plant sterols-enriched soya beverage for consecutive 3 weeks, each pack consumed once with main meal (i.e breakfast, lunch or dinner).
  Plant sterols-enriched soya beverage: the study product is a 2g plant sterols-enriched in 250ml soya beverage
- Soya Beverage: Daily consumption of one pack of 250 ml of soya beverage (without plant sterols) for consecutive 3 weeks, each pack consumed once with main meal (i.e breakfast, lunch or dinner).
  Soya beverage: the placebo product is a 250 ml soya beverage
Arm/Group | Plant Sterols-enriched Soya Beverage | Soya Beverage
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/101
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/101
Other Adverse Events (participants affected / at risk) | 5/100 | 1/101
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Plant Sterols-enriched Soya Beverage (N=100) | Soya Beverage (N=101)
Diarrhea (Gastrointestinal disorders) | 3 | 0
Stomach Bloating (Gastrointestinal disorders) | 0 | 1
Slight hardening of stool during the three weeks period (Gastrointestinal disorders) | 1 | 0
Flu (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-17): https://cdn.clinicaltrials.gov/large-docs/58/NCT02881658/Prot_SAP_000.pdf